CLINICAL TRIAL: NCT01147601
Title: Topical Timolol 0.5% Solution for Proliferating Infantile Hemangiomas: A Prospective Double Blinded Placebo Controlled Study
Brief Title: Topical Timolol 0.5% Solution for Proliferating Infantile Hemangiomas
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Dr. Alfons Krol, MD, FRCPC, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6114
Record Dates: First submitted 2010-06-14; First posted 2010-06-22 (Estimated); Results first posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-04

CONDITIONS: Hemangioma; Infant
Keywords: topical 0.5% Timolol; infantile hemangioma (IH)
MeSH Terms: conditions — Hemangioma; Hemangioma, Capillary | interventions — Timolol; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical 0.5% Timolol (Active Comparator): Half of the enrolled subjects (intervention group) will receive topical 0.5% Timolol.
  Interventions: Drug: topical 0.5% Timolol
- Placebo (Placebo Comparator): Aqueous placebo, 2-3 drops to cover the hemangioma, twice daily
  Interventions: Drug: Control (placebo) group

INTERVENTIONS:
Drug: topical 0.5% Timolol — topical 0.5% Timolol aqueous solution, 2-3 drops to cover the hemangioma, twice daily
  Arms: Topical 0.5% Timolol
Drug: Control (placebo) group — Control (placebo) group
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn about a new potential use for topical timolol 0.5% aqueous solution that may help treat small uncomplicated infantile hemangiomas. This study would examine whether topical timolol could be a potential therapy.

DETAILED DESCRIPTION:
At the first visit, subjects will fill out a questionnaire that asks about the child's history and the hemangioma. Photographs and measurements will be taken at this and each subsequent visit. At the first visit, subjects will have a physical exam, including vital signs, height and weight. An EKG will also be done. Study drug will be dispensed and instructions given. Half of the subjects will receive a placebo. This is a blinded randomized study. Follow-up visits will be weekly for the first two weeks (three visits total including the first visit), then monthly until the study is over. Photographs and measurements will again be taken at each visit. Subjects will be asked to evaluate the size and the color of the hemangioma against the first photographs and fill out forms regarding any changes in behavior and asked about any side effects.

ELIGIBILITY:
Inclusion Criteria:

Infants 1 month to 8 months of age with infantile hemangioma (IH) that are 3 cm or less on the scalp, trunk, or extremities.

Exclusion Criteria:

1. Subjects with facial, genital, perianal, hand, finger, feet, or toe IH
2. Subjects with PHACES (plaque-like hemangioma on the face awaiting imaging) syndrome (proven) or suspected PHACES .
3. Subjects with IH measuring more than 3cm in size or ulcerated.
4. Children with a history of hypersensitivity to beta blockers.
5. Children with a personal history of asthma.
6. Children with known renal impairment.
7. Children with known cardiac conditions that may predispose to heart block
8. Personal history of hypoglycemia
9. Children on medications that may interact with beta blockers

Ages: 1 Month to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2010-03; Primary Completion 2012-10 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfons L. Krol, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topical 0.5% Timolol | Placebo
Started | 5 | 1
Completed | 2 | 1
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical 0.5% Timolol | Placebo | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Continuous [Mean (Full Range); unit: days] | 93.5 [41 to 217] | 178 [178 to 178] | 123.2 [41 to 217]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects in Treatment Group Compared to Placebo Group With at Least 75% Improvement in the Extent of the Hemangioma as Compared to Baseline Photos.
Description: This will be generated by asking each of the assessors to score the improvement using a visual analog scale (VAS) assessing the decrease in size of hemangioma by comparing photographs at different times of treatment. The assessors will score this improvement into one of the following categories: 0-24%, 25-49%, 50-74%, >75%.
Time Frame: at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Topical 0.5% Timolol | Placebo
Number analyzed (Participants) | 2 | 1
Participants | 1 | 0

2. Secondary Outcome: Compare Treatment Group to Control Group Improvement Assessments
Description: 1. The proportion of subjects in the treatment group as compared to the placebo control group with at least 50% improvement in the extent of the hemangioma.
  2. The difference between the extent/size of the hemangioma as an outcome measure versus color changes.
  3. Frequency of adverse events (e.g. hypotension, behavioral changes, etc.), collected by the investigator and reported by the parents.
Time Frame: at 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Topical 0.5% Timolol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/1
Other Adverse Events (participants affected / at risk) | 1/5 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical 0.5% Timolol (N=5) | Placebo (N=1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes